CLINICAL TRIAL: NCT01008215
Title: Cluster Randomized Trial to Assess the Effect of Using a Simple Warfarin Maintenance Dosing Algorithm on the Quality of INR Control Among Canadian Family Practices
Brief Title: Simple Warfarin Dosing Algorithm Study
Acronym: KT-INR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Dr. Stuart Connolly, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-282
Record Dates: First submitted 2009-10-28; First posted 2009-11-05 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Warfarin Dosing
Keywords: INR Control; Warfarin dosing; Family physicians; Cluster randomization
MeSH Terms: interventions — Algorithms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Algorithm (Experimental): Algorithm (available in paper version and web-based version) will be used for warfarin maintenance dosing.
  Interventions: Other: Algorithm
- Care as usual (No Intervention): Control group

INTERVENTIONS:
Other: Algorithm — Warfarin Dosing algorithm (paper and electronic version)
  Arms: Algorithm

SUMMARY:
Can a simple and cost-free tool help family physicians to improve dosing of the blood thinner warfarin?

Warfarin is a blood thinner with a variable effect and requires regular blood monitoring and dose adjustments. Some family practices do not have the facilities or funding to use commercial tools than can assist with stabilizing the effect of warfarin. The investigators will test whether a simple and cost-free dosing tool can help these practices to improve warfarin management.

If this simple tool improves warfarin management, it will be freely available for practices in Canada and around the world. This will help physicians who have no access to more costly and/or complicated tools improve their warfarin dosing practice in a systematic fashion, and thereby maximize the health benefit of warfarin.

DETAILED DESCRIPTION:
Warfarin reduces the risk of thromboembolism, but requires regular blood monitoring to keep the international normalized ration (INR) within a narrow therapeutic range to achieve maximum benefits. A low proportion of time spent within the therapeutic INR range, (TTR) is associated with reduced warfarin efficacy and potentially harmful results. To optimize TTR, international guidelines recommend the use of systematic evidence-based dosing methods (anticoagulation clinic, computerized systems, manual algorithm and patient self-management). A survey in the Hamilton area revealed that half of family physicians manage warfarin dosing without assistance from an evidence-based method. The simple manual dosing algorithm is a simple tool that helped increase the TTR at the Hamilton General Hospital's anticoagulant clinic to an excellent 73% among patients with target INR range 2-3. We will test whether the simple dosing algorithm can help to improve warfarin dosing of family physicians who are not assisted by evidence-based methods. We will randomize family practices to either use the simple dosing algorithm or to manage warfarin dosing as usual, to test whether the simple dosing algorithm achieves a superior TTR.

ELIGIBILITY:
Inclusion Criteria:

* Family practices that:

  1. currently do not employ an evidence-based dosing method (anticoagulant clinic, computer system, manual algorithm or patient self-testing),
  2. manage warfarin maintenance dosing in at least 10 patients with target INR 2-3, and
  3. have at least one family physician providing written informed consent.
* Patients who:

  1. are on long-term warfarin treatment (> 6 weeks before study entry and expected to continue for at least 6 more months) with target INR 2-3, for whom warfarin is managed by a participating family physician,
  2. patient provides written informed consent.

Exclusion Criteria:

* Family practices that:

  1. are planning to start employing an evidence-based method for warfarin dosing within the next year,
  2. are not expected to enroll at least 10 patients on long-term warfarin treatment with target INR 2-3.
* Patients:

  1. with < 3 months warfarin management prior to the baseline observation,
  2. patients on warfarin with a target INR other than 2-3, and
  3. patients for whom warfarin is managed by a physician who is not participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mean time in therapeutic range for patients | 1 Year

SECONDARY OUTCOMES:
Proportion of patients with TTR > 65% | 1 Year
Correlation between algorithm adherence and TTR | 1 Year
Among patients in both baseline and study sample: proportion of patients with TTR improvement | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, Principal Investigator — McMaster University
Locations (1):
- Caroline Medical Group, Burlington, Ontario, Canada